CLINICAL TRIAL: NCT02890823
Title: EFFECT OF THREE DIFFERENT DOSES OF ORAL CHOLECALCIFEROL (1000 IU, 3000 IU AND 6000 IU DAILY) ON SERUM 25-HYDROXYVITAMIN D CHANGES AMONG EPILEPSY PATIENTS WITH HYPOVITAMINOSIS D: A RANDOMIZED PROSPECTIVE STUDY
Brief Title: Effect of Three Different Doses of Oral Cholecalciferol on 25-Hydroxyvitamin D Changes Among Epilepsy Patients With Hypovitaminosis D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA58/075
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Epilepsy
Keywords: Antiepileptic Drugs; Vitamin D Deficiency; Asian
MeSH Terms: conditions — Epilepsy; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- EIAEDs-1000 (Experimental): Patients receiving EIAEDs who were randomly assigned to receive vitamin D3 1000 IU once daily
  Interventions: Drug: Cholecalciferol
- EIAEDs-3000 (Experimental): Patients receiving EIAEDs who were randomly assigned to receive vitamin D3 3000 IU once daily
  Interventions: Drug: Cholecalciferol
- EIAEDs-6000 (Experimental): Patients receiving EIAEDs who were randomly assigned to receive vitamin D3 6000 IU once daily
  Interventions: Drug: Cholecalciferol
- non-EIAEDs-1000 (Active Comparator): Patients receiving non-EIAEDs who were randomly assigned to receive vitamin D3 1000 IU once daily
  Interventions: Drug: Cholecalciferol
- non-EIAEDs-3000 (Active Comparator): Patients receiving non-EIAEDs who were randomly assigned to receive vitamin D3 3000 IU once daily
  Interventions: Drug: Cholecalciferol
- non-EIAEDs-6000 (Active Comparator): Patients receiving non-EIAEDs who were randomly assigned to receive vitamin D3 6000 IU once daily
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol

SUMMARY:
To characterize the effect of three different doses of vitamin D3 supplementation on serum 25-hydroxyvitamin D (25(OH)D) changes in epilepsy patients receiving enzyme-inducing antiepileptic drugs (EIAEDs) versus patients receiving non enzyme-inducing antiepileptic drugs (non-EIAEDs), and to determine the prevalence of and risk factors for hypovitaminosis D among Thai patients with epilepsy.

DETAILED DESCRIPTION:
A single-blinded prospective, randomized study undertaken at epilepsy clinic of King Chulalongkorn Memorial Hospital. The patients with hypovitaminosis D were included and divided into two groups according to the type of AEDs use. Patients receiving each AEDs type were randomly assigned to receive vitamin D3 1000, 3000 or 6000 IU once daily. The mean increment in serum 25(OH)D levels were measured at 8 and 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy patients, age ≥ 15 years, BMI18 - 30 kg/m2
* Being treated with either enzyme inducing antiepileptic drugs (EIAEDs: phenytoin, phenobarbital, carbamazepine and topiramate) or non-enzyme inducing antiepileptic drugs (Non-EIAEDs: sodium valproate, levetiracetam, and lamotrigine) at a stable dosage regimen for at least a year.
* Serum 25(OH)D <30ng/ml

Exclusion Criteria:

* Patients with a history of hypercalcemia, nephrolithiasis, fractures, hepatic disease, kidney disease, granulomatous disease or currently supplemented with vitamin D.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
serum 25-hydroxyvitamin D changes in patients who received enzyme-inducing antiepileptic drugs (EIAEDs) versus patients receiving non enzyme-inducing antiepileptic drugs (non-EIAEDs) at the same dosage of cholecalciferal | 8 and 16 months

SECONDARY OUTCOMES:
Number (percentage) of the patients who have serum 25-hydroxyvitamin D levels more than 30ng/ml | 16 months